CLINICAL TRIAL: NCT05046158
Title: Randomized Clinical Trial to Compare Transforming Powder and Standard of Care Dressing Therapies to Heal Diabetic Foot Ulcers
Brief Title: Diabetic Foot Ulcers-Comparing Transforming Powder to Standard of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ULURU Inc. (Industry)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Military Technology Enterprise Consortium (US) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-C-TPD-2021-01
Record Dates: First submitted 2021-08-17; First posted 2021-09-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: Standard of Care Wound Dressings; Transforming Powder Dressing; Diabetic Foot Ulcers; Altrazeal
MeSH Terms: conditions — Diabetic Foot | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: Randomized, Prospective, Multi-Center, Open-Label, Comparison, Human, Interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transforming Powder Dressing (Active Comparator): Half of the subjects will be randomized to Transforming Powder Dressing to treat their diabetic foot ulcers. Wounds will be evaluated weekly, debrided if needed, photographed, and measured. A wound dressing will be applied using Transforming Powder Dressing and the wound will be offloaded when necessary (pressure taken off of the wound using a total contact cast or other device). Wound healing progress will be monitored and compared to other standard of care dressings used to treat diabetic foot ulcers.Surveys regarding pain and quality of life will be completed at each study visit.
  Interventions: Device: Transforming Powder Dressing
- Standard of Care Dressing (Active Comparator): Half of the subjects will be randomized to receive standard of care wound dressings to treat their diabetic foot ulcers. Wounds will be evaluated weekly, debrided if needed, photographed, and measured. A wound dressing will be applied using standard of care wound products, and the wound will be offloaded when necessary (pressure taken off of the wound using a total contact cast or other device). Wound healing progress will be monitored and compared to transforming powder dressings used to treat diabetic foot ulcers. Surveys regarding pain and quality of life will be completed at each study visit.
  Interventions: Other: Standard of care topical wound agents and dressings

INTERVENTIONS:
Device: Transforming Powder Dressing — Altrazeal transforming powder dressing is methacrylate-based powder dressing made from the same materials used in the production of contact lenses. Upon hydration, the powder transforms into a moist, non-occlusive barrier that covers and protects the wound from exogenous bacteria while helping manage exudate through vapor transpiration.
  Other Names: Altrazeal
  Arms: Transforming Powder Dressing
Other: Standard of care topical wound agents and dressings — Standard wound dressings such as gauze or foams. Moisture regulating topical agents may also be used to prepare the wound bed.
  Arms: Standard of Care Dressing

SUMMARY:
Phase IV, randomized, prospective, multi-center, open-label, comparison of transforming powder dressing to standard of care dressing for healing diabetic foot ulcers.

DETAILED DESCRIPTION:
Diabetic men and women aged 18-89 years, who have a diabetic foot ulcer present for a minimum of 30 days will be considered for the study. Subjects will be randomized to either standard of care wound dressings or transforming powder dressing. Half of the subjects will receive standard of care dressings, and the other half will receive transforming powder dressing in a 1:1 randomization process at each of the study sites. Subjects will present to the study center weekly for up to 12 weeks (less time if the wound heals prior to 12 weeks). The last study visit occurs 12 weeks after the End of Study visit.

ELIGIBILITY:
Inclusion Criteria:

* 18-89 years old
* Diagnosed with diabetes Mellitus; hemoglobin A1C < 12%
* Diabetic foot ulcer present for minimum 30 days (Wagner grade 1 or 2 classification)
* Wound drainage is minimal or moderate
* No clinically active wound infection
* Able and willing to provide consent
* Has not participated in another research trial within 3 months of enrollment.

Exclusion Criteria:

* Unable to keep weekly research appointments
* Unable or unwilling to use offloading device if recommended
* Wounds with large amount (high) drainage
* Active gangrene
* Wounds impending surgical intervention (including revascularization or plastic surgery)
* Untreated osteomyelitis
* Soft tissue infection (can be enrolled once infection is cleared)
* Active Charcot arthropathy
* BMI >45kg/m2
* History of AIDS
* History of organ transplant or impending transplant
* End stage renal disease requiring dialysis
* Decompensated hepatic or cardiac disease
* Select autoimmune diseases
* Lymphedema
* Oral steroid use in last 3 months
* Venous stasis disease
* Active malignancy (cancer)
* Unable to sign consent
* Active alcohol or substance abuse
* Pregnant or lactating women
* Insufficient vascular flow to heal a wound
* Hemoglobin A1C >12%

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Incidence of wound closure | 12 weeks
  Compare rate of complete wound healing in diabetic foot wounds between the two study groups

SECONDARY OUTCOMES:
Wound healing trajectories and time to wound closure | 12 weeks
  Evaluate differences in wound healing trajectories and time to wound closure between the two study groups
Adverse Events | 12 weeks
  Safety as indicated by adverse events (new or worsening conditions) and frequency of wound infections
Subject Satisfaction | 12 weeks
  Evaluate subject satisfaction of wound care products based on "Research subject satisfaction survey" completed at the end of study (8 questions total using a 7 point Likert scale).
Wound pain | 12 weeks
  Compare differences in pain between the groups based on results of a validated 10 point "Visual Analogue Pain Scale" completed at each visit by all subjects. More pain is indicated by higher scores.
Quality of Life while living with a wound | 12 weeks
  Compare differences in quality of life between the groups based on results of completed validated "Wound Quality of Life Questionnaire for Chronic Wounds" (17 questions total, answering a 5 point scale [not at all to very much], results from answers based on formula)
Clinician Acceptability | 12 weeks
  Based on clinician survey completed at end of study (8 questions total, multiple choice or 7 point Likert scale)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM, MPH, Principal Investigator — Altrazeal Life Sciences Inc.; Jonathan Saxe, MD, Study Director — Altrazeal Life Sciences Inc.
Locations (12):
- United States (12):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Medical Group Foot & Ankle at Winter Park, Winter Park, Florida
  - VA Maryland Health Care System, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - MedStar Franklin Square, Rossville, Maryland
  - Northwell Health Wound Healing Center, Lake Success, New York
  - Bronx Foot Care, The Bronx, New York
  - James J. Peters VA Medical Center, The Bronx, New York
  - VA Hudson Valley HealthCare System, Wappingers Falls, New York
  - Dallas Veteran's Administration Medical Center, Dallas, Texas
  - Baylor College of Medicine Clinic Hospital McNair (MDHP) BCM390, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schaper NC, van Netten JJ, Apelqvist J, Bus SA, Hinchliffe RJ, Lipsky BA; IWGDF Editorial Board. Practical Guidelines on the prevention and management of diabetic foot disease (IWGDF 2019 update). Diabetes Metab Res Rev. 2020 Mar;36 Suppl 1:e3266. doi: 10.1002/dmrr.3266. PMID 32176447
- [Background] Han G, Ceilley R. Chronic Wound Healing: A Review of Current Management and Treatments. Adv Ther. 2017 Mar;34(3):599-610. doi: 10.1007/s12325-017-0478-y. Epub 2017 Jan 21. PMID 28108895
- [Background] Wound Care Awareness Week Highlights of the Chronic Wound Epidemic in U.S. Businesswire.com/news/home/20160607006326/en/Wound-Care-Awareness-Week-Highlights-Chronic-Wound. Accessed 11/5/2020.
- See also: Altrazeal (Transforming Powder Dressing) product information — http://www.Altrazeal.info